CLINICAL TRIAL: NCT04171700
Title: A Phase 2 Multicenter, Open-label Study of Rucaparib as Treatment for Solid Tumors Associated With Deleterious Mutations in Homologous Recombination Repair Genes
Brief Title: A Study to Evaluate Rucaparib in Participants With Solid Tumors and With Deleterious Mutations in HRR Genes
Acronym: LODESTAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to a change in development priorities.
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-100
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor
Keywords: rucaparib; PARPi; rare tumor; solid tumor; CO-338; ovarian cancer; prostate cancer; pancreatic cancer; breast cancer; lung cancer; colon cancer; gastric cancer; bladder cancer; colorectal cancer; PARP inhibitor; homologous recombination; DNA repair; LODESTAR; germline; somatic; BRCA1; BRCA2; PALB2; RAD51C; RAD51D; BARD1; BRIP1; FANCA; RAD51; RAD51B; sarcoma; HRR; HRD; platinum sensitive; platinum resistant; primary peritoneal cancer; fallopian tube cancer; tumor agnostic; basket study; basket trial; metastatic; locally advanced; esophageal cancer; leiomyosarcoma; ampullary carcinoma; carcinosarcoma; endometrial cancer; cervical cancer
MeSH Terms: conditions — Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms; Sarcoma; Fallopian Tube Neoplasms; Neoplasm Metastasis; Esophageal Neoplasms; Leiomyosarcoma; Carcinosarcoma; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib (Experimental): Eligible participants will be enrolled in either Cohort A or Cohort B.
  Cohort A: Up to 200 participants with deleterious mutations in BRCA1, BRCA2, PALB2, RAD51C or RAD51D.
  Cohort B (Exploratory): Up to 20 participants with deleterious mutations in BARD1, BRIP1, FANCA, NBN, RAD51 or RAD51B.
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Oral rucaparib will be administered twice daily. The starting dose will be 600 mg daily (BID).
  Other Names: Rubraca; Rucaparib camsylate; Rucaparib tablets; CO-338; PF 01367338; AG 014447

SUMMARY:
A Phase 2, open-label, single-arm trial to evaluate the response of rucaparib in participants with various solid tumors and with deleterious mutations in Homologous Recombination Repair (HRR) genes.

ELIGIBILITY:
Key Inclusion Criteria:

* Unresectable, locally advanced or metastatic solid tumor and relapsed/progressive disease
* Measurable disease per RECIST v1.1 or modified RECIST v1.1 and PCWG3 (for prostate cancer)
* Have a deleterious mutation (germline or somatic) in BRCA1, BRCA2, PALB2, RAD51C, RAD51D, BARD1, BRIP1, FANCA, NBN, RAD51 or RAD51B. Note: Breast cancer patients that are HER2 negative and have germline BRCA1 or BRCA2 mutations AND patients with epithelial ovarian cancer, fallopian tube cancer, primary peritoneal cancer or metastatic castration-resistant prostate cancer with BRCA1 or BRCA2 mutations are ineligible for this trial.
* At least one prior line of therapy extending overall survival or standard of care therapy for advanced disease. Note: Some tumor types have specific inclusion/exclusion criteria for previous treatments.
* ECOG 0 or 1
* Tumor tissue available for genomic analysis, or must be willing to have a biopsy if no archival tumor tissue available
* Adequate organ function
* Life expectancy of 4 months

Key Exclusion Criteria:

* Active central nervous system brain metastases, leptomeningeal disease or primary tumor of CNS origin
* Active second malignancy (Exceptions: Successfully treated malignancy with no active disease for 1 year, surgically cured and/or low-risk tumors, or patients receiving ongoing anticancer hormonal therapy for a previously treated cancer)
* Pre-existing gastrointestinal disorders/conditions interfering with ingestion/absorption of rucaparib
* Prior treatment with a PARP inhibitor
* More than 3 prior lines of chemotherapy in the locally advanced/metastatic setting
* History of myelodysplastic syndrome or acute myeloid leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Reiss-Binder, MD, Principal Investigator — University of Pennsylvania
Locations (19):
- United States (19):
  - UCLA Medicine Hematology and Oncology, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Beth Israel Deaconess Medical Cancer Surgical Pavilion, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - New York Cancer And Blood Specialists, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center - The University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI/Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Seattle Cancer Care Alliance/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets for study results will be made available to qualified researchers in compliance with applicable privacy laws and data protection regulations.
  Data will be provided by Clovis Oncology.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to qualified researchers after the primary, secondary, and/or exploratory outcomes of the study are reported or published and for 1 year thereafter.
Access Criteria: Requests for de-identified datasets will be made available to qualified researchers following submission of a methodologically sound proposal to medinfo@clovisoncology.com.

REFERENCES:
- [Derived] Anbil S, Seewald NJ, Chiorean EG, Hussein M, Kasi PM, Laux DE, Schwartz GK, Shapiro GI, Lin KK, Craib M, Maloney L, McLachlan K, Tukachinsky H, Schrock AB, Wang S, Sokol ES, Decker B, Nathanson KL, Domchek SM, Reiss KA. LODESTAR: A Single-Arm Phase II Study of Rucaparib in Solid Tumors With Pathogenic Germline or Somatic Variants in Homologous Recombination Repair Genes. JCO Precis Oncol. 2025 Jul;9:e2500090. doi: 10.1200/PO-25-00090. Epub 2025 Jul 9. PMID 40632975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 83 participants were enrolled across 19 US sites between January 2020 and March 2022. 63 participants were enrolled in cohort A and 20 in cohort B.
  Cohort A comprised participants with a deleterious mutation in one of the following genes; BRCA1, BRCA2, PALB2, RAD51C, RAD51D.
  Cohort B comprised participants with a deleterious mutation in one of the following genes: BARD1, BRIP1, FANCA, NBN, RAD51, RAD51B.
Groups:
- Rucaparib Cohort A: Participants with a deleterious mutation in one of the following genes: BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.
- Rucaparib Cohort B: Participants with a deleterious mutation in one of the following genes: BARD1, BRIP1, FANCA, NBN, RAD51, or RAD51B.
Period: Overall Study
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Started | 63 | 20
Completed | 63 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B | Total
Number analyzed (Participants) | 63 | 20 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 8 | 41
  >=65 years | 30 | 12 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (10.85) | 65.2 (13.38) | 64.8 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 14 | 50
  Male | 27 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 61 | 20 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 56 | 19 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 20 | 83

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate by Investigator
Description: Best overall response rate as assessed by the investigator by RECIST v1.1 (or by RECIST v1.1 and PCWG3 in participants with advanced prostate cancer).
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: Efficacy population - all participants evaluable for response by RECIST v1.1 (or modified RECIST v1.1/PCWG3 for mCRPC participants).
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 61 | 20
Participants | 9 | 2

2. Secondary Outcome: Overall Response Rate by Independent Radiology Review
Description: Best overall response rate by independent radiology review by RECIST v1.1 (or by RECIST v1.1 and PCWG3 in participants with advanced prostate cancer).
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: No data were collected as the independent radiology review was not performed.
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of Response
Description: Measure of clinical benefit, defined as the time from initial tumor response to documented tumor progression.
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Rucaparib Cohort B: Participants with a deleterious mutation in one of the following genes: BRD1, BRIP1, FANCA, NBN, RAD51, or RAD51B.
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 9 | 2
month | 4.1 [3.1 to NA] — Insufficient number of participants with events. | 6.8 [2.6 to 10.9]

4. Secondary Outcome: Disease Control Rate
Description: Measure of clinical benefit, defined as the percentage of complete response (CR), partial response (PR), and stable disease (SD) beyond 16 weeks.
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 61 | 20
percentage of participants | 36.1 [24.2 to 49.4] | 25.0 [8.7 to 49.1]

5. Secondary Outcome: Progression-free Survival
Description: Measure of clinical benefit, defined as the duration from study enrollment to objective tumor progression. Progression was defined using RECIST v1.1, as a 20% increase in the sum of diameters of target lesions (and an absolute increase of at least 5 mm), or unequivocal progression of existing non-target lesions, or the appearance of new lesions. For mCRPC disease, the PCWG3 confirmed bone disease progression criteria (2+2) were also incorporated.
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: Safety Population - all enrolled participants who received at least 1 dose of protocol-specified treatment.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 63 | 20
month | 3.7 [1.9 to 5.4] | 3.6 [1.6 to 6.3]

6. Secondary Outcome: Overall Survival
Description: Measure of clinical benefit, defined as the duration from study enrollment to death.
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: Safety Population - all enrolled participants who received at least 1 dose of protocol-specified treatment.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 63 | 20
month | 13.3 [10.6 to NA] — Insufficient number of participants with events. | 8.0 [4.8 to 16.6]

7. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: Safety Population - all enrolled participants who received at least 1 dose of protocol-specified treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 63 | 20
Participants | 63 | 20

8. Secondary Outcome: Steady State Minimum Concentration [Cmin]
Description: Rucaparib pharmacokinetics
Time Frame: From first dose of study drug until disease progression (up to approximately 2 years)
Population: Pharmacokinetics data not collected due to early study termination.
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of first dose of study drug until 28 days after the last dose of study drug, approximately 2 years.
Description: Adverse events are reported for the Safety Population, defined as participants who received at least one dose of protocol-specified treatment.
Arm/Group | Rucaparib Cohort A | Rucaparib Cohort B
All-Cause Mortality (participants affected / at risk) | 23/63 | 10/20
Serious Adverse Events (participants affected / at risk) | 13/63 | 5/20
Other Adverse Events (participants affected / at risk) | 63/63 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib Cohort A (N=63) | Rucaparib Cohort B (N=20)
Anemia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib Cohort A (N=63) | Rucaparib Cohort B (N=20)
Anemia (Blood and lymphatic system disorders) | 20 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 23 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 25 | 8
Stomatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 18 | 5
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 31 | 10
Oedema peripheral (General disorders) | 6 | 2
Pyrexia (General disorders) | 6 | 0
COVID-19 (Infections and infestations) | 5 | 0
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 7 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Alanine aminotransferase increased (Investigations) | 10 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Blood cholesterol increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 7 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 0
International normalized ratio increased (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 8 | 0
Neutrophil count decreased (Investigations) | 10 | 2
Platelet count decreased (Investigations) | 7 | 3
Weight decreased (Investigations) | 6 | 1
Weight increased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 10 | 1
Decreased appetite (Metabolism and nutrition disorders) | 15 | 4
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 7 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 1
Hyponatremia (Metabolism and nutrition disorders) | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 11 | 1
Dysguesia (Nervous system disorders) | 8 | 5
Headache (Nervous system disorders) | 6 | 3
Lethargy (Nervous system disorders) | 3 | 1
Tremor (Nervous system disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Chromaturia (Renal and urinary disorders) | 2 | 1
Hematuria (Renal and urinary disorders) | 4 | 1
Proteinuria (Renal and urinary disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04171700/Prot_SAP_001.pdf